### **Statistical Analysis Plan (SAP)**

# A Prospective, Multi-Center Evaluation of a Powered Vascular Stapler in Video-Assisted Thoracoscopic Lobectomies

**Protocol Number: ESC-14-006** 

Protocol Version: Original, February 11, 2016

This document is a confidential communication. The recipient agrees that no unpublished information contained herein will be published or disclosed without prior written approval. This document may be disclosed to the appropriate ethics committees or to duly authorized representatives of the U.S. Food and Drug Administration or other responsible regulatory authorities, under the condition that they are requested to keep it confidential.

**SAP Revision:** 1.0 **SAP Revision Date:** 06JUL2017

# **Revision History**

| Revision Number | Revision Date | Reasons for Revision |
|-----------------|---------------|----------------------|
| 1.0 | 06JUL2017 | Original Document |

### **Table of Contents**

| 1 | Study Overview | . 4 |
|-------|----------------------------------------------------------|-----|
| | 1.1 Study Objectives | 4 |
| | 1.2 Study Design | 4 |
| 2 | Treatment Assignment | 4 |
| 3 | Randomization and Blinding Procedures | 4 |
| 4 | Interval Windows | 4 |
| 5 | Primary and Secondary Endpoints | . 5 |
| | 5.1 Primary Effectiveness Endpoint | . 5 |
| | 5.2 Primary Safety Endpoint | . 5 |
| | 5.3 Secondary and Additional Endpoints | . 5 |
| 6 | Levels of Significance | . 5 |
| 7 | Analysis Sets | 6 |
| 8 | Sample Size Justification | 6 |
| 9 | Data Monitoring Committee (DMC) | 6 |
| 10 | Analyses to be Conducted | . 7 |
| | 10.1 General Conventions | . 7 |
| | 10.2 Disposition of Study Subjects | . 7 |
| | 10.3 Demographic, Baseline, and Surgical Characteristics | . 7 |
| | 10.4 Primary Endpoint Analyses | . 7 |
| | 10.5 Plans for Interim Analysis | 9 |
| | 10.6 Handling of Missing Data | 9 |
| | 10.7 Sensitivity Analyses | 9 |
| | 10.8 Subgroup Analysis | 9 |
| | 10.9 Assessment of Site Homogeneity | 9 |
| | 10.10 Additional Endpoint Analyses | 9 |
| | 10.11 Safety Analyses | 10 |
| Appen | ndix: Table Shells and List of Listings to be Generated | 10 |

This is the Statistical Analysis Plan (SAP) for the final analysis of data collected under Protocol ESC-14-006. This SAP describes in detail the statistical methodology and statistical analyses for the above mentioned protocol.

# 1 Study Overview

## 1.1 Study Objectives

The primary objective was to demonstrate the effectiveness of the powered vascular stapler (PVS) for transection of the pulmonary artery (PA) and pulmonary vein (PV) during video-assisted thoracoscopic surgery (VATS) lobectomy.

### 1.2 Study Design

This was a prospective, multi-center study that collected data from the surgeon's use of the PVS for PA/PV transection. Prospective subjects were informed about the nature of the research, given the ICD to read, and if the subject understood the consent, was asked to provide written consent (the ICD).

# 2 Treatment Assignment

This was a single-arm study where all enrolled subjects underwent VATS lobectomy with the planned usage of PVS for transection of the PA and PV.

# 3 Randomization and Blinding Procedures

This was a single-arm, open-label study. No randomization occurred and no blinding procedures were required.

### 4 Interval Windows

Interval windows are not defined for the purpose of analysis in this study as the collection of data for the primary performance endpoint occurred intra-operatively and the collection of data for the primary safety endpoint occurred through hospital discharge. The final visit occurred approximately 4 weeks after surgery, thus no interval windows need to be defined given the absence of long-term follow-up in this study. The study protocol specified a window of 5 days around the scheduling of the 4-week follow-up visit, and any information entered in the eCRFs at this visit will correspond to the 4-week visit. There will be no assigning of observations to time points outside of the visit to which they are recorded in the eCRFs. The complete Schedule of Events for this study can be found in the Synopsis of the study protocol.

# 5 Primary and Secondary Endpoints

### 5.1 Primary Effectiveness Endpoint

The primary effectiveness endpoint in this study was defined as the occurrence of hemostatic interventions/procedures completed for intra-operative bleeding related to the transection of the PA and PV during VATS lobectomy. Hemostasis interventions or procedures were defined as bleeding detected and controlled intra-operatively (additional stapling, over-sewing, clip placement, compression, use of suture, sealant, and/or buttress, and/or use of energy); or bleeding that occurred intra-operatively requiring blood or blood product transfusion or an additional surgical procedure (e.g. conversion to open). No hemostasis intervention was defined as no bleeding at the staple line or bleeding that stopped after initial blotting of the staple line.

The primary effectiveness endpoint will be summarized at the firing level as multiple firings per subject were expected and observed; that is, the denominator for the primary endpoint will be the total number of firings and the numerator will be the number of firings where an intervention was required.

### 5.2 Primary Safety Endpoint

The primary safety endpoint was defined as the occurrence of hemostatic interventions/procedures completed for post-operative bleeding related to the transection of the PA and PV during VATS lobectomy. Hemostasis intervention was defined as bleeding that occurred post-operatively requiring blood or blood product transfusion or an additional surgical procedure (related to PA and PV transection). No hemostasis intervention was defined as no interventions needed for post-operative bleeding (related to PA and PV transection). This endpoint was recorded at the subject level as it was based on post-operative interventions and not specific to any individual firing.

### 5.3 Secondary and Additional Endpoints

Key additional endpoints in this study include: pain score assessments, American Shoulder and Elbow Surgeons Standardized (ASES) Shoulder Assessment, Surgeon Task Load Index, adverse events, and device usability questionnaires.

# 6 Levels of Significance

No hypotheses are specified for this study and no p-values are being calculated, therefore no level of significance is specified. All estimation of endpoints will be performed using 95% confidence intervals.

# 7 Analysis Sets

There will be three analysis sets defined:

- The Full Analysis Set (FAS) will consist of all enrolled subjects who had a procedure completed and provided data on the number of surgical interventions;
- The Per Protocol (PP) Analysis Set will consist of all subjects in the FAS who had no major protocol deviations. Determination of major deviations are conducted by the study Medical Director, Project Manager and Biostatistician. A major deviation is defined as: A departure from the study protocol that has the potential to affect the scientific validity of the study (including deviations that: a) impact the analysis of the primary endpoint, or b) are due to inappropriate enrollment of a subject that does not meet the inclusion/exclusion criteria) or the safety, rights and welfare of the enrolled subject.
- The Safety Analysis Set will consist of all enrolled subjects on whom a procedure was started.

The primary effectiveness endpoint analysis will be performed on the Full Analysis Set. The primary effectiveness endpoint analysis will also be performed on the PP set as a sensitivity analysis to the results on the FAS. A summary of additional endpoints will also be performed on the Full Analysis Set. Analysis of the primary safety endpoint and adverse events summaries will be performed on the Safety Analysis Set.

# 8 Sample Size Justification

Approximately 50 subjects were enrolled in the study. No formal sample sizing was performed for this study as it is a single-arm study without a hypothesis. Historical clinical study data on a similar powered surgical stapler demonstrated a need for staple line interventions in approximately 6% of firings on the pulmonary artery or pulmonary vein. This data also showed an average of 2.6 to 2.9 firings per subject, and it is expected, given differences in device design, that each subject will require 3 to 4 firings on the pulmonary vein or pulmonary artery in the current study with PVS. Therefore, assuming an average of 3.5 firings per subject, a sample size of 50 subjects should provide approximately 175 firings. Assuming a 6% proportion of firings which require an intra-operative hemostatic intervention/procedure background rate, then the proposed sample size should control the margin of error for a 95% confidence interval to be no more than 3.5% and provide adequate precision for evaluating the performance of PVS and allow for qualitative comparisons to additional trials involving this device.

# 9 Data Monitoring Committee (DMC)

No Data Monitoring Committee was planned or utilized during this study.

# 10 Analyses to be Conducted

### 10.1 General Conventions

Subject data will be summarized using listings and tables. All eCRF data will be listed per subject for all subjects. Descriptive statistical analyses will be provided for pre-specified study endpoints. Summaries for continuous variables will include number of observations (n), mean, standard deviation, median, minimum, and maximum. Summaries for categorical variables will include number and percentage.

Analyses will be conducted using SAS software version 9.4 or higher. During the course of analysis programming of tables that are mocked up in this SAP, minor modifications may become necessary. Examples of these minor modifications include, but are not limited to, re-wording of a footnote, addition of a footnote, re-labeling of a column, or addition or removal of a column from a listing. In cases where modifications to tables or listings are not related to a change in statistical analysis methodology or conclusions that could be made on the originally proposed methodology, then no amendment of the SAP is necessary. Any final analyses that differ from what has been specified in this document will be identified within the final statistical output and documented within the clinical study report.

### 10.2 Disposition of Study Subjects

Subject disposition will be summarized in total using counts and percentages. The number and percentage of subjects in each analysis set will be tabulated. Additionally, the number and percentage of subjects completed and discontinued will be tabulated along with the specific reasons for discontinuation.

### 10.3 Demographic, Baseline, and Surgical Characteristics

Summary statistics of subject demographics (age, gender, race, and ethnicity) will be presented in total for the Full Analysis Set. Surgical characteristics including, at minimum, lobe location, calcified hilar lymph node presence, number of ports used, number of pulmonary arteries transected, number of chest tubes placed, ASA physical status, estimated blood loss, conversion to open, requirement for blood transfusion, procedure duration, and number of chest tubes will be summarized in total. Results of tumor assessments performed by the pathology laboratory (including tumor stage, maximum tumor diameter, maximum tumor depth, primary TNM classification, presence of distant metastasis, and confirmation of non-small cell lung cancer) will also be summarized.

### 10.4 Primary Endpoint Analyses

For the primary performance endpoint, summary statistics and a 95% confidence interval will be provided for the number and percentage of interventions for the FAS. To account for the potential dependence among firings within a subject, the 95% confidence interval will be estimated using a

bootstrap approach. For each subject, the outcome of each firing will be represented by a vector of 0's (indicating no intervention needed) and 1's (indicating an intervention was needed). This vector will be re-sampled with replacement to generate a bootstrap sampled vector of observations for each subject. Then, the proportion of observations requiring intervention for each subject will be calculated from this bootstrap vector. After obtaining a sample proportion of firings requiring intervention for each subject, the mean of these sample proportions will be calculated across all 50 subjects to provide an estimated sample proportion of firings requiring intervention based on 1 iteration of the bootstrap process. This process will then be repeated a minimum of 5000 times to generate a sampling distribution for the proportion of firings requiring intervention. The mean of this sampling distribution will be provided as the point estimate of the proportion of firings requiring intervention and the 95% confidence interval will be estimated by the lower 0.025 and upper 0.975 percentiles of this sampling distribution.

The table below demonstrates 1 iteration of this bootstrap process.

| Subject | Observed Data Vector | Bootstrap Sampled | Bootstrap-Based Sample |
|---|---|---|---|
| ID | | Vector | Proportion |
| 1 | (0, 0, 1, 0, 0) | (0, 1, 0, 1, 0) | 0.40 |
| 2 | (0,0,0) | (0,0,0) | 0.0 |
| 3 | (0, 1, 0, 0) | (1, 0, 0, 0) | 0.25 |
| 4 | (0, 0, 1, 0, 0) | (0, 0, 0, 0, 0) | 0.0 |
| 5 | (0,0) | (0,0) | 0.0 |
| 50 | (1, 0, 0, 1, 0) | (0, 1, 0, 0, 0) | 0.20 |
| Summary | | | Average of above proportions |
| | | | to get 1 observation in the |
| | | | sampling distribution of the |
| | | | proportion of firings requiring |
| | | | intervention. |

The above re-sampling process will then be repeated a minimum of 5000 times to estimate the sampling distribution.

A secondary estimate of the proportion of firings requiring intervention will be provided under the assumption of independence of firings within a subject. This will be performed based on the total number of firings and the percentage will be calculated as the number of firings requiring an intervention divided by the total number of firings. The 95% confidence interval will be estimated using exact Binomial methods.

Additional summaries will be provided to tabulate the total number of vessels transected as well as the specific type of vessel that was transected – pulmonary artery or pulmonary vein. The specific types of interventions that were performed will also be tabulated.

The same analysis will be replicated for the primary safety endpoint for the occurrence of hemostatic interventions/procedures completed for post-operative bleeding related to the transection of the PA and PV during VATS lobectomy at the subject level. Here, the percentage will be calculated as the number of subjects requiring a post-operative intervention divided by the total number of subjects. The 95% confidence interval will be estimated using exact Binomial methods.

### 10.5 Plans for Interim Analysis

No interim analyses were planned or performed for this study.

### 10.6 Handling of Missing Data

All summaries will be performed only on subjects undergoing the VATS procedure and only observed data will be summarized. There will be no imputation of data for early terminated subjects or for missing data within the database.

### 10.7 Sensitivity Analyses

Analyses of the primary effectiveness and safety endpoints will be replicated on the Per Protocol Set to assess the primary results in the set of subjects with no major protocol violations. Exploratory analyses of the primary endpoint data will be performed where measurements within a subject are assumed to be correlated. Given the smaller sample size of this study, data from this protocol may be combined with data from Protocol ESC-15-001 to allow for a more robust analysis. Binomial models utilizing generalized estimating equations to account for repeated measures within a subject will be applied to the data to estimate whether correlation exists and to provide estimates for the rate of interventions as a sensitivity analysis to the primary results.

### 10.8 Subgroup Analysis

No subgroup analyses are planned for this study.

### 10.9 Assessment of Site Homogeneity

No summaries or adjustments by study site are planned for this study.

### 10.10 Additional Endpoint Analyses

Device usage details will be summarized with counts and percentages for subjects in whom the device was articulated during the surgical procedure. Similar summaries will also be provided for the surgeon satisfaction questionnaire and the surgeon device questionnaire.

Post-operative pain is assessed at Visit 3 and Visit 4. Subjects are asked to rate their pain on a scale ranging from 0 (no pain) to 10 (worst possible pain). Subjects will rate pain relating to three sites – trocar site, incisional site, and chest tube site. Summary statistics at each pain site will be provided at Visits 3 and 4, as well as the change from Visit 3 to Visit 4.

Summary statistics will be provided for the Surgery Task Load Index (Surg-TLX). Surgeons are asked to rate 6 specific components after each surgery performed. The 6 components are – mental fatigue, physical fatigue, hurried/rushed pace, procedure complexity, anxious while performing procedure, and distracting operating environment. Each component is scored on a 0 to 100 scale with lower scores representing a 'Low' response on that component and higher scores indicating a 'High' response on that component. Summaries will also be provided for an overall score which is calculated as the average of the six components for each surgery.

The ASES Shoulder Assessment is a patient reported outcome designed to measure functional limitations and pain of the shoulder and has been adapted to this study to measure upper body functionality following VATS lobectomy. The assessment utilizes 10 questions that are answered with: unable to do = 0, very difficult to do = 1, somewhat difficult to do = 2, and not difficult = 3. Scores for each subject are obtained by summing the responses to the 10 questions and thus range from 0 to 30. Summary statistics will be provided for the ASES Shoulder Assessment at Visit 1 (prior to surgery), Visit 3 (after surgery, prior to discharge), and Visit 4 (approximately 4 weeks after surgery). Summary statistics will also be provided for the change from Visit 1 to Visit 3, and for the change from Visit 1 to Visit 4.

The total number of protocol deviations will be tabulated. Specific types of protocol deviations will also be summarized with counts and percentages. The number and percentage of subjects with at least one protocol deviation will also be summarized.

### 10.11 Safety Analyses

Safety will be assessed through the incidence of adverse events (AEs) and serious adverse events (SAEs), which will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). The number and percentage of subjects reporting AEs and SAEs will be summarized at the MedDRA system organ class and preferred term level. Similar summaries will also be provided for AEs and SAEs related to the study device, as well as for AEs and SAEs related to the study procedure. Related events are those where the relationship is indicated as Possibly, Related, or Unknown. The incidence of AEs will also be summarized by maximum severity. All reported adverse events will be listed.

# Appendix: Table Shells and List of Listings to be Generated

Table shells are provided below for all summaries to be generated for this study. Additionally, a list of all listings to be created is provided corresponding to the eCRFs that were used during this study. All fields collected will be listed.

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm


Table 1 Subject Disposition All Subjects

| | Total |
|-----------------------------|------------|
| Signed Informed Consent | XX |
| Safety Set | xx (xx.x%) |
| Full Analysis Set | xx (xx.x%) |
| Completed the Study | xx (xx.x%) |
| Discontinued from the Study | xx (xx.x%) |
| Leason for Discontinuation | |
| Withdrawal of consent | xx (xx.x%) |
| Surgical | xx (xx.x%) |
| Adverse Event | xx (xx.x%) |
| Death | xx (xx.x%) |
| Lost to Follow-up | xx (xx.x%) |
| Site or Study Termination | xx (xx.x%) |
| Other | xx (xx.x%) |

Note: All percentages are based on the number of subjects in the Safety Set as the denominator.

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 2 Subject Demographics Full Analysis Set

| Characteristics | Overall (N = ##) |
|-------------------------------------------|------------------|
| | (2 ,) |
| Race | |
| White | xx (xx.x%) |
| Black or African American | xx (xx.x%) |
| American Indian or Alaska Native | xx (xx.x%) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x%) |
| Asian | xx (xx.x%) |
| Other | xx (xx.x%) |
| Ethnicity | |
| Han | xx (xx.x%) |
| Other | xx (xx.x%) |
| Subject did not want to disclose | xx (xx.x%) |
| Age (years) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Gender | |
| Male | xx (xx.x%) |
| Female | xx (xx.x%) |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 3 Protocol Deviations Safety Set

| Characteristics | Overall (N = ##) |
|---|---|
| Total Number of Protocol Deviations | xxx |
| Specific Types of Protocol Deviations [1] | |
| Informed Consent Process | xx (xx.x%) |
| Inclusion/Exclusion Criteria | xx (xx.x%) |
| Study Procedure | xx (xx.x%) |
| Visit Out of Window | xx (xx.x%) |
| Other | xx (xx.x%) |
| Sponsor Assessment of Protocol Deviations [1] | |
| Minor | xx (xx.x%) |
| Major | xx (xx.x%) |
| Number (%) of Subjects With at Least 1 Protocol Deviation [2] | xx (xx.x%) |

 Ethicon Inc. Protocol: ESC-14-006

SAP Version 1.0: 06JUL2017

Denominator used is the total number of protocol deviations reported.
 Denominator used is the total number of subjects in the column header.

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4 Surgical Characteristics Full Analysis Set

| Characteristics | Overall<br>(N = ##) |
|-----------------------------------------------|--------------------------|
| X | |
| Location of Affected Lobe | (0/) |
| Left Lung, Superior Lobe | xx (xx.x%) |
| Left Lung, Inferior Lobe | xx (xx.x%) |
| Left Lung, Multiple Lobes | xx (xx.x%) |
| Right Lung, Superior Lobe | xx (xx.x%) |
| Right Lung, Middle Lobe | xx (xx.x%) |
| Right Lung, Inferior Lobes | xx (xx.x%) |
| Right Lung, Multiple Lobes | xx (xx.x%) |
| Calcified Hilar Lymph Nodes Present? | |
| Yes | xx(xx.x%) |
| No | xx (xx.x%) |
| Number of Pulmonary Arteries Transected | |
| 0 | xx (xx.x%) |
| 1 | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| NI L CD 4 | |
| Number of Ports | (0/) |
| 1 | xx (xx.x%) |
| 2 | xx (xx.x%) |
| 3 | xx (xx.x%) |
| 4 | xx (xx.x%) |
| Number of Chest Tubes Placed Intraoperatively | |
| 0 | xx (xx.x%) |
| 1 | xx (xx.x%) |
| 2 | xx (xx.x%) |
| ASA Physical Status | |
| Class I | xx (xx.x%) |
| Class II | xx (xx.x%) |
| Class III | xx (xx.x%)<br>xx (xx.x%) |
| C1055 111 | AX (AX.A/0) |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 4 Surgical Characteristics Full Analysis Set

| | Overall |
|-------------------------------------------------|---------------|
| Characteristics | (N = ##) |
| Characteristics | (11 "") |
| Estimated Blood Loss (mL) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Transfusion of Blood or Blood Product Required? | 6.00 |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Procedure Converted to Open? | |
| Yes | xx(xx.x%) |
| No | xx (xx.x%) |
| Procedure Duration (min) | |
| n | XX |
| Mean | XX X |
| Standard Deviation | XX.X<br>X.XXX |
| Median | XX.X |
| Minimum, Maximum | |
| Millingin, Maximum | XX.X, XX.X |
| Chest Tube Duration (nights) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |

Programming Note: Chest tube duration is calculated from date of surgery to date of final chest tube removal

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 5 Tumor Assessment – Pathology Lab Full Analysis Set

| | Overall |
|-------------------------------------|--------------------------|
| Characteristics | (N = ##) |
| Tumor Stage, Confirmed by Pathology | |
| Stage 0 | xx (xx.x%) |
| Stage IA | xx (xx.x%) |
| Stage IB | xx (xx.x%) |
| Stage IIA | xx (xx.x%) |
| Stage IIA<br>Stage IIB | xx (xx.x%) |
| Stage IIIA | xx (xx.x%) |
| Stage IIIA<br>Stage IIIB | xx (xx.x%)<br>xx (xx.x%) |
| Stage IIIB<br>Stage IV | |
| Stage IV | xx (xx.x%) |
| Maximum Tumor Diameter (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Maximum Tumor Depth (cm) | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | x.xxx |
| Median | XX.X |
| Minimum, Maximum | XX.X, XX.X |
| Primary Tumor TNM Classification | |
| TX | xx (xx.x%) |
| TO | XX (XX.X%) |
| Tix | xx (xx.x%) |
| T1 | xx (xx.x%) |
| Tla | xx (xx.x%) |
| Tlb | xx (xx.x%) |
| T2 | xx (xx.x%) |
| T3 | xx (xx.x%) |
| T4 | xx (xx.x%)<br>xx (xx.x%) |

Ethicon Inc. Protocol: ESC-14-006 SAP Version 1.0: 06JUL2017 

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm
Data Last Modified: mm/dd/yyyy hh:mm

Table 5 Tumor Assessment – Pathology Lab Full Analysis Set

| Characteristics | Overall<br>(N = ##) |
|---|---|
| TNM Classification for Regional Lymph Node | |
| NX | xx(xx.x%) |
| N0 | xx (xx.x%) |
| N1 | xx (xx.x%) |
| N2 | xx (xx.x%) |
| N3 | xx (xx.x%) |
| Distant Metastasis Present? | |
| Yes | xx(xx.x%) |
| No | xx (xx.x%) |
| Tumor Confirmed by Pathology as Non-Small Cell Lung Cancer? | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |

Ethicon Inc. Protocol: ESC-14-006 SAP Version 1.0: 06JUL2017 

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm


Table 6 Intra-Operative Interventions on Pulmonary Artery or Pulmonary Vein Full Analysis Set

| Characteristics | Overall (N = ##) |
|---|---|
| | , , |
| Total Number of Vessels Transected | XXX |
| Pulmonary Artery | XXX |
| Pulmonary Vein | XXX |
| Bootstrap Based Summary Statistics | |
| Bootstrap Mean | xx.x% |
| 95% Confidence Interval from Bootstrap Sampling Distribution | XX.X%, XX.X% |
| Number of Vessel Transections Requiring Intervention [1] | |
| n (%) | xx (xx,x%) |
| 95% Confidence Interval for Percent | XX.X%, XX.X% |
| Type of Intervention, n (%) [2] | |
| Additional Stapling | xx (xx,x%) |
| Over-sewing | xx (xx.x%) |
| Compression | xx (xx.x%) |
| Use of Suture | xx (xx.x%) |
| Sealant | xx (xx.x%) |
| Buttress | xx (xx.x%) |
| Use of Energy | xx (xx.x%) |
| Clip Placement | xx (xx.x%) |
| Blood Product Transfusion | xx (xx.x%)<br>xx (xx.x%) |
| Additional Surgical Procedure | xx (xx.x%)<br>xx (xx.x%) |
| Other Intervention | xx (xx.x%) |
| outer intervention | AA (AA.A/0) |

<sup>[1]</sup> Denominator for calculation of percentage is the total number of vessels transected. Confidence interval based on exact Binomial method.

<sup>[2]</sup> Denominator for calculation of percentage is the total number of vessels requiring intervention.

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 7 Post-Operative Interventions or Procedures Related to Pulmonary Artery or Pulmonary Vein Bleeding Safety Set

| Characteristics | Overall (N = ##) |
|---|---|
| Number of Subjects Requiring Post-Operative Intervention Related | |
| to Pulmonary Artery or Pulmonary Vein Bleeding | |
| n (%) [1] | xx (xx.x%) |
| 95% Confidence Interval for Percent | xx.x%, xx.x% |
| Type of Intervention, n (%) [2] | |
| Blood Product Transfusion | xx (xx.x%) |
| Additional Surgical Procedure | xx (xx.x%) |
| Other Intervention | xx (xx.x%) |

Ethicon Inc. Protocol: ESC-14-006 

SAP Version 1.0: 06JUL2017

<sup>[1]</sup> Denominator for calculation of percentage is the total number of subjects in that group.
[2] Denominator for calculation of percentage is the total number of subjects requiring intervention in that group.

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 8 Device Usage Details Full Analysis Set

| Characteristics | Overall (N = ##) |
|---|---|
| Number of Subjects Where Device Was Articulated | xxx |
| Did Articulation Make it Easier to Perform Surgery? [1]<br>Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Was Articulation Essential to Performing the Surgery? [1] | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |
| Was the Angle Range of the Device Sufficient? [1] | |
| Yes | xx (xx.x%) |
| No | xx (xx.x%) |

<sup>1.</sup> Denominator used is the total number of subjects in whom the device was articulated.

Ethicon Inc. Protocol: ESC-14-006 

SAP Version 1.0: 06JUL2017

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 9 Surgery Task Load Index (SURG-TLX) Full Analysis Set

| Characteristic | Overall (N = ##) |
|---|---|
| | , |
| Overall Score | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Mentally Fatiguing | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Physically Fatiguing | |
| n | XX |
| Mean | XX.X |
| Standard Deviation | X.XXX |
| Median | XX.X |
| Minimum, Maximum | xx.x, xx.x |
| Similar summaries for remaining components:<br>Hurried/Rushed Pace<br>Procedure Complexity<br>Anxious While Performing Procedure<br>Distracting Operating Environment | |

Note: Each component is scored on a 0 to 100 scale with lower scores representing a 'Low' response and higher scores representing a 'High' response.

Ethicon Inc. Protocol: ESC-14-006 SAP Version 1.0: 06JUL2017 

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm
Data Last Modified: mm/dd/yyyy hh:mm

Table 10 Surgeon Satisfaction Questionnaire Full Analysis Set

| Characteristics | Overall (N = ##) |
|---------------------------------------------|------------------|
| How Satisfied Were You With Device Usabilit | v? |
| Very Unsatisfied | xx (xx.x%) |
| Unsatisfied | xx (xx.x%) |
| Neutral | xx (xx.x%) |
| Satisfied | xx (xx.x%) |
| Very Satisfied | xx (xx.x%) |
| Amount of Tissue Slippage | |
| No Tissue Slippage | xx (xx.x%) |
| Some Tissue Slippage | xx (xx.x%) |
| Extensive Tissue Slippage | xx (xx.x%) |

Ethicon Inc. Protocol: ESC-14-006 SAP Version 1.0: 06JUL2017 

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 11 Post-Operative Pain Score Full Analysis Set

| Pain Component | Time Point<br>Statistic | Overall (N = ##) |
|----------------|--------------------------------|------------------|
| Tam Component | Statistic | (14 ##) |
| Trocar Pain | Visit 3 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | x.xxx |
| | Median | XX.X |
| | Minimum, Maximum | xx.x, xx.x |
| | Visit 4 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| | Change From Visit 3 to Visit 4 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |

Same summary will be repeated for:

Incisional Pain Chest Tube Pain

Programming note: Change from Visit 3 to Visit 4 will be calculated as Visit 4 value minus Visit 3 value.

Note: For each pain component, the subject is asked to rate his or her pain today on a scale from 0 (no pain) to 10 (worst possible pain).

Ethicon Inc. Protocol: ESC-14-006 

SAP Version 1.0: 06JUL2017

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

### Table 12 Surgeon Device Questionnaire Full Analysis Set

| Question | Overall |
|---|---|
| Response | (N = ##) |
| The ECHELON FLEX Powered Vascular Stapler with Advanced Placement Tip enables | |
| easier placement of the device on vessels compared to your current standard of care device: | |
| Strongly Disagree | xx (xx.x%) |
| Slightly Disagree | xx (xx.x%) |
| Neutral | xx (xx.x%) |
| Agree | xx (xx.x%) |
| Strongly Agree | xx (xx.x%) |
| The ECHELON FLEX Powered Vascular Stapler with Advanced Placement Tip has the | |
| potential to reduce the amount of dissection required (otomy) around the vessel to place the | |
| stapler compared to your current standard of care device: | |
| Strongly Disagree | xx (xx.x%) |
| Slightly Disagree | xx (xx.x%) |
| Neutral | xx (xx.x%) |
| Agree | xx (xx.x%) |
| Strongly Agree | xx (xx.x%) |
| The ECHELON FLEX Powered Vascular Stapler with Advanced Placement Tip has the potential to reduce the surgeon stress during the most challenging step of the procedure, which is the pulmonary artery / pulmonary vein transection, compared to your current standard of care device: | 1 |
| Strongly Disagree | xx (xx.x%) |
| Slightly Disagree | xx (xx.x%) |
| Neutral | xx (xx.x%) |
| Agree | xx (xx.x%) |
| Strongly Agree | xx (xx.x%) |
| The ECHELON FLEX Powered Vascular Stapler with Advanced Placement Tip allows for the precise control and placement of the end effector on the target vessel compared to your current standard of care device: | |
| Strongly Disagree | xx (xx.x%) |
| Slightly Disagree | xx (xx.x%)<br>xx (xx.x%) |
| Neutral | xx (xx.x%)<br>xx (xx.x%) |
| Agree | xx (xx.x%) |
| Strongly Agree | xx (xx.x%) |
| buongry rigivo | AA (AA.A/0) |

Ethicon Inc. Protocol: ESC-14-006 SAP Version 1.0: 06JUL2017 

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 13 ASES Shoulder Assessment Full Analysis Set

| | Time Point | Overall |
|---------------|--------------------------------|------------|
| Shoulder Side | Statistic | (N = ##) |
| B. 1. | *** | |
| Right | Visit 1 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| | Visit 3 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| | Change From Visit 1 to Visit 3 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| | Visit 4 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |
| | Change From Visit 1 to Visit 4 | |
| | n | XX |
| | Mean | XX.X |
| | Standard Deviation | X.XXX |
| | Median | XX.X |
| | Minimum, Maximum | XX.X, XX.X |

Same summary will be repeated for: Left Side

Programming note: Change from Visit 1 to Visit 3 will be calculated as Visit 3 value minus Visit 1 value.

 Ethicon Inc. Protocol: ESC-14-006

SAP Version 1.0: 06JUL2017

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 14 Adverse Events by System Organ Class and Preferred Term Safety Set

| System Organ Class | Preferred Term | Overall<br>(N = ##) |
|---|---|---|
| Total | | xx (xx.x%) |
| System Organ Class 1 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 2 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 3 | Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| System Organ Class 4 | Preferred Term 1<br>Preferred Term 2 | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following tables will have the same format as Table 14:

| Table 15 | Serious Adverse Events by System Organ Class and Preferred Term |
|---|---|
| | Safety Set |
| Table 16 | Adverse Events Related to the Study Device by System Organ Class and Preferred Term |
| | Safety Set |
| Table 17 | Serious Adverse Events Related to the Study Device by System Organ Class and Preferred Term |
| | Safety Set |
| Table 18 | Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term |
| | Safety Set |
| Table 19 | Serious Adverse Events Related to the Study Procedure by System Organ Class and Preferred Term |
| | Safety Set |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

Table 20 Adverse Events by System Organ Class, Preferred Term and Maximum Severity Safety Set

| System Organ Class | Preferred Term | Overall (N = ##) |
|----------------------|------------------|------------------|
| System Organ Class | Treferred Term | (11 ##) |
| Total | | xx (xx.x%) |
| Mild | | xx (xx.x%) |
| Moderate | | xx (xx.x%) |
| Severe | | xx (xx.x%) |
| System Organ Class 1 | | xx (xx.x%) |
| Mild | | xx (xx.x%) |
| Moderate | | xx (xx.x%) |
| Severe | | xx (xx.x%) |
| | Preferred Term 1 | xx (xx.x%) |
| | Mild | xx (xx.x%) |
| | Moderate | xx (xx.x%) |
| | Severe | xx (xx.x%) |
| | Preferred Term 2 | xx (xx.x%) |
| | Mild | xx (xx.x%) |
| | Moderate | xx (xx.x%) |
| | Severe | xx (xx.x%) |
| System Organ Class 2 | | xx (xx.x%) |
| Mild | | xx (xx.x%) |
| Moderate | | xx (xx.x%) |
| Severe | | xx (xx.x%) |
| | Preferred Term 1 | xx (xx.x%) |
| | Mild | xx (xx.x%) |
| | Moderate | xx (xx.x%) |
| | Severe | xx (xx.x%) |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm

The following listings will be generated for this study:

| Listing 1 | Inclusion/Exclusion Criteria |
|---|---|
| | All Subjects |
| Listing 2 | Demographics |
| | All Subjects |
| Listing 3 | Medical History |
| | All Subjects |
| Listing 4 | Surgical History |
| | All Subjects |
| Listing 5 | Inclusion/Exclusion at Surgery and ASA Status |
| | All Subjects |
| Listing 6 | Procedure Details |
| | All Subjects |
| Listing 7 | Procedure Time Duration |
| | All Subjects |
| Listing 8 | Intra-Operative Interventions on Pulmonary Artery and Pulmonary Vein |
| | All Subjects |
| Listing 9 | Bronchus and Parenchyma Transections |
| | All Subjects |
| Listing 10 | Intra-Operative Interventions Not on Pulmonary Artery and Pulmonary Vein |
| | All Subjects |
| Listing 11 | Device Usage Details |
| | All Subjects |
| Listing 12 | Tumor Assessment Log |
| | All Subjects |
| Listing 13 | Surgeon Device Questionnaire |
| | All Subjects |
| Listing 14 | Surgery Task Load Index |
| | All Subjects |
| Listing 15 | Surgeon Satisfaction Questionnaire |
| | All Subjects |

Protocol Number: ESC-14-006

Page x of y

Program Name: XXXXXXXX.sas Run Date: mm/dd/yyyy hh:mm Data Last Modified: mm/dd/yyyy hh:mm


| Listing 16 | Post-Operative Interventions on Pulmonary Artery and Pulmonary Vein All Subjects |
|---|---|
| Listing 17 | Pain Score Assessment All Subjects |
| Listing 18 | Chest Tube Details Log<br>All Subjects |
| Listing 19 | Adverse Events All Subjects |
| Listing 20 | Concomitant Medications All Subjects |
| Listing 21 | Concomitant Procedures/Interventions All Subjects |
| Listing 22 | Protocol Deviations All Subjects |
| Listing 23 | Completion/Withdrawal All Subjects |
| Listing 24 | Study Visits All Subjects |